CLINICAL TRIAL: NCT03099109
Title: A Phase 1a/1b Study of LY3321367, an Anti-TIM-3 Antibody, Administered Alone or in Combination With LY3300054, an Anti-PD-L1 Antibody, in Advanced Relapsed/Refractory Solid Tumors
Brief Title: A Study of LY3321367 Alone or With LY3300054 in Participants With Advanced Relapsed/Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16526; I9A-MC-JLDA (Other: Eli Lilly and Company); 2016-003195-42 (EudraCT Number)
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor
Keywords: TIM-3; PD-L1
MeSH Terms: interventions — LY3321367; LY3300054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- LY3321367 Dose Escalation (Experimental): LY3321367 given intravenously (IV).
  Interventions: Drug: LY3321367
- LY3321367 + LY3300054 Dose Escalation (Experimental): LY3321367 and LY3300054 given IV.
  Interventions: Drug: LY3321367; Drug: LY3300054
- LY3321367 Dose Expansion (Experimental): LY3321367 given IV.
  Interventions: Drug: LY3321367
- LY3321367 + LY3300054 Dose Expansion (Experimental): LY3321367 and LY3300054 given IV.
  Interventions: Drug: LY3321367; Drug: LY3300054
- Japanese Arm D LY3321367 (Experimental): LY3321367 given IV.
  Interventions: Drug: LY3321367
- Japanese Arm E LY3300054 (Experimental): LY3300054 given IV.
  Interventions: Drug: LY3300054
- Japanese Arm F LY3321367 + LY3300054 (Experimental): LY3321367 and LY3300054 given IV.
  Interventions: Drug: LY3321367; Drug: LY3300054

INTERVENTIONS:
Drug: LY3321367 — Administered IV
  Arms: Japanese Arm D LY3321367; Japanese Arm F LY3321367 + LY3300054; LY3321367 + LY3300054 Dose Escalation; LY3321367 + LY3300054 Dose Expansion; LY3321367 Dose Escalation; LY3321367 Dose Expansion
Drug: LY3300054 — Administered IV
  Arms: Japanese Arm E LY3300054; Japanese Arm F LY3321367 + LY3300054; LY3321367 + LY3300054 Dose Escalation; LY3321367 + LY3300054 Dose Expansion

SUMMARY:
The purpose of this study is to evaluate the safety of the study drug known as LY3321367, an anti-T-cell immunoglobulin and mucin-domain domain-containing molecule-3 (TIM-3) antibody administered alone or in combination with LY3300054, an anti-programmed death ligand 1 (PD-L1) antibody, in participants with advanced relapsed/refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* For Ph1a monotherapy and combination cohorts, histologic or cytologic confirmation of advanced solid tumor.
* For Phase 1a and 1b, prior PD-1 or PD-L1 therapy or other immunotherapy is allowed, if the following criteria are met:

  * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
  * Must have completely recovered or recovered to baseline prior to screening from any prior AEs occurring while receiving prior immunotherapy.
* Must have provided tumor tissue sample, as follows:

  * For participants entering Ph1a: have submitted, if available, an archival tumor tissue sample.
  * For participants entering Ph1b: have submitted, a sample from a newly obtained core or excisional biopsy of a tumor lesion or a recent biopsy defined by 6 months of study enrollment (Ph1b).
* Must have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Must have adequate organ function.
* Have an estimated life expectancy of 12 weeks, in judgement of the investigator.

Exclusion Criteria:

* Have symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids (participants receiving anticonvulsants are eligible).
* Have received a live vaccine within 30 days before the first dose of study treatment.
* If female, is pregnant, breastfeeding, or planning to become pregnant.
* Have a history or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the participant's participation.
* Have moderate or severe cardiovascular disease.
* Have a serious concomitant systemic disorder that would compromise the participant's ability to adhere to the protocol, including active or chronic infection with human immunodeficiency virus (HIV), active hepatitis B virus (HBV), active hepatitis C virus (HCV), active autoimmune disorders, or prior documented severe autoimmune or inflammatory disorders requiring immunosuppressive treatment.
* Use of escalating or chronic supraphysiologic doses of corticosteroids or immunosuppressive agents (such as, cyclosporine). [Use of topical, ophthalmic, inhaled, and intranasal corticosteroids permitted].
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection.
* Evidence of interstitial lung disease or noninfectious pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with DLTs | Baseline through Cycle 1 (28 Day Cycle)
  Dose Limiting Toxicity (DLT) is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.

SECONDARY OUTCOMES:
PK: Cmax of LY3321367 | Cycle 1 Day 1 through Follow-Up (Estimated up to 6 Months)
  Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3321367
PK: Cmax of LY3321367 in Combination with LY3300054 | Cycle 1 Day 1 through Follow-Up (Estimated up to 6 Months)
  Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3321367 in Combination with LY3300054
ORR: Percentage of Participants With a CR or PR | Baseline to Measured Progressive Disease (Estimated up to 6 Months)
  Objective Response Rate (ORR) is the percentage of participants with confirmed best overall tumor response of Complete Response (CR) or Partial Response (PR).
PFS | Baseline to Objective Progression or Death Due to Any Cause (Estimated Up to 12 Months)
  Progression Free Survival (PFS) is defined as the date of the first dose to the first date of objectively determined progressive disease or death from any cause, whichever is earlier.
DoR | Date of CR or PR to Date of Objective Progression or Death Due to Any Cause (Estimated up to 12 Months)
  Duration of Response (DoR) is defined as the time from the date of the first CR or PR to the first date of progressive disease (PD) or death from any cause.
TTR | Baseline to Date of CR or PR (Estimated up to 6 Months)
  Time to Response (TTR) is defined as time from treatment start to first documentation of response.
DCR: Percentage of Participants who Exhibit SD, CR or PR | Baseline through Measured Progressive Disease (Estimated up to 6 Months)
  Disease Control Rate (DCR) is the percentage of participants with stable disease (SD), confirmed PR or confirmed CR (CR+PR+SD).

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM- 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (8):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University College of Phys & Surgeons, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Peggy and Charles Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The START Center for Cancer Care, San Antonio, Texas
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (3):
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Fundación Jiménez Díaz-Oncology, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid

REFERENCES:
- [Derived] Harding JJ, Moreno V, Bang YJ, Hong MH, Patnaik A, Trigo J, Szpurka AM, Yamamoto N, Doi T, Fu S, Calderon B, Velez de Mendizabal N, Calvo E, Yu D, Gandhi L, Liu ZT, Galvao VR, Leow CC, de Miguel MJ. Blocking TIM-3 in Treatment-refractory Advanced Solid Tumors: A Phase Ia/b Study of LY3321367 with or without an Anti-PD-L1 Antibody. Clin Cancer Res. 2021 Apr 15;27(8):2168-2178. doi: 10.1158/1078-0432.CCR-20-4405. Epub 2021 Jan 29. PMID 33514524
- See also: A Study of LY3321367 Alone or With LY3300054 in Participants With Advanced Relapsed/Refractory Solid Tumors — https://www.lillytrialguide.com/en-US/studies/solid-tumor/JLDA#?postal=